CLINICAL TRIAL: NCT04384601
Title: Efficacy Study of FLOT Versus SOX Regimen as Neoadjuvant Chemotherapy for Patients With Locally Advanced Gastric Cancer: A Phase 3 Multi-center Randomized Controlled Trial
Brief Title: Dragon III-Phase 3: Neoadjuvant Chemotherapy (FLOT Versus SOX) for Gastric Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BIRENDRA KUMAR SAH, Surgeon, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dragon III-Phase 3
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer; Neoadjuvant Chemotherapy
Keywords: Gastric Cancer; Gastric Adenocarcinoma; Stomach Cancer, Adenocarcinoma; Chemotherapy Effect; Neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOX Chemotherapy (Experimental): Three preoperative and three postoperative cycles of SOX chemotherapy
  A cycle consist of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil potassium capsule 80mg/M2 oral (twice daily)
  Repeated every 21st day
  Interventions: Drug: Chemotherapy
- FLOT Chemotherapy (Active Comparator): Four preoperative and four postoperative cycles of FLOT chemotherapy
  A cycle consist of Day 1 5-fluorouracil(5-FU) 2600mg/M2 administered via intravenous peripherally inserted central venous catheter(PICC) for 24 hour Leucovorin 200mg/M2 intravenous Oxaliplatin 85mg/ M2 intravenous Docetaxel 50mg/M2 intravenous
  Repeated every 15th day
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Perioperative chemotherapy will be administered according to description in two arms.
  Other Names: FLOT chemotherapy; SOX chemotherapy

SUMMARY:
DRAGON III research, Neoadjuvant Chemotherapy (FLOT versus SOX) for Gastric Cancer, is an investigator initiated; phase 3, open label, multi-center randomized controlled study.

DETAILED DESCRIPTION:
Non inferiority of SOX will be tested against FLOT. This study will be conducted at multiple center of China and will invite international centers to join it.The sponsor of this study is Ruijin Hospital and the project is supported by the Shanghai Key Laboratory of Gastric Neoplasms and Institute of Digestive Surgery, Shanghai.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed non-obstructive adenocarcinoma of stomach or esophago-gastric junction.
* Clinical stage: Clinical Tumor-Node-Metastasis (cTNM:) stage III
* Performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2 (normal to symptomatic but in bed less than half the day)
* Clinically fit for systemic chemotherapy and gastric cancer surgery, i.e. adequate renal, hepatic, hematologic and pulmonary function.
* Written informed consent

Exclusion Criteria:

* Clinically unfit for systemic chemotherapy and gastric cancer surgery, i.e. uncontrolled cardiac disease, or other clinically significant uncontrolled comorbidities, unable to undergo general anesthesia
* Distant metastases (including retroperitoneal lymph node)
* Locally advanced inoperable disease (Clinical assessment)
* Relapse of gastric cancer
* Malignant secondary disease
* Prior chemo or radio therapy
* Inclusion in another clinical trial
* Known contraindications or hypersensitivity for planned chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total Percentage of Patients With Pathological Complete Tumor Regression (TRG1a) and Sub-total Tumor Regression (TRG1b) in the Primary Tumour | Upto three months
  Tumor regression grade (TRG), Becker criteria Grade 1a :Complete tumor regression: 0% residual tumor per tumor bed Grade 1b: Subtotal tumor regression: <10% residual tumor per tumor bed Grade 2: Partial tumor regression: 10-50% residual tumor per tumor bed Grade 3: Minimal or no tumor regression: >50% residual tumor per tumor bed

SECONDARY OUTCOMES:
Overall Survival (OS) | Five years
  Overall survival Time from randomization to death from any cause
Disease free survival (DFS) | Three years
  Disease free survival Time from randomization to relapse or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Birendra K Sah, PH D, Principal Investigator — Ruijin Hospital; Chen Li, PH D, Study Director — Ruijin Hospital; Zhenggang Zhu, PH D, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No